CLINICAL TRIAL: NCT03264183
Title: Validating Transesophageal Echocardiographic Measurements of Right Ventricular Function
Brief Title: Validating TEE Measurements of Right Ventricular Function
Acronym: TEE
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Shayne Michael Roberts, Assistant Professor, Milton S. Hershey Medical Center
Other Study IDs: STUDY00007541
Record Dates: First submitted 2017-07-26; First posted 2017-08-29 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Ventricular Function, Right; Echocardiography, Transesophageal
MeSH Terms: interventions — Echocardiography, Transesophageal; Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography — TEE measures of right ventricular function
  Other Names: TEE
Diagnostic Test: Transthoracic Echocardiography — TTE measures of right ventricular function
  Other Names: TTE

SUMMARY:
Transesophageal echocardiography (TEE) is becoming a more prevalent method of monitoring and diagnosis in the perioperative setting for critically ill patients and patients undergoing cardiac surgery. Many TEE measurements are extrapolated from transthoracic echocardiography (TTE) data and have not validated by transesophageal means. The aim of this study is to validate TEE assessment of right ventricular function by comparing them to simultaneously measured TTE measurements.

Likewise, there are currently no agreed upon values for RV free wall strain. Therefore, the investigators will attempt to define a range of normal values of RV free wall strain as compared to the other measures of RV function.

DETAILED DESCRIPTION:
Traditionally, all echocardiographic measurements have been studied utilizing TTE. Therefore the normal values and ranges for pathology findings have been defined by transthoracic means alone. TEE offers different images planes when compared to TTE, which may make the measurements obtained differ from those obtained by TTE. In the operating room environment the vast majority of echocardiography is completed by transesophageal means for many reasons; largely access to the patient and the continuous use of TEE as a hemodynamic monitor. However, given the fact that most echocardiographic measurements have only been validated by TTE, there remains a question as to the validity or precision of TEE-derived measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective cardiac surgery requiring TEE

Exclusion Criteria:

* Patient who do not wish to consent
* Patients with contraindications to TEE
* Urgent or emergent cardiac surgery
* Patients with preexisting open chest
* Patients with intrathoracic hardware (VAD, thoracostomy tube, etc)
* Non-English speaking subjects
* Cognitively impaired adults
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective cardiac surgery, which as a standard of care, requires transesophageal echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Right ventricular index of myocardial performance (RIMP) | Immediately following the induction of anesthesia and TEE probe placement
  Right ventricular index of myocardial performance (RIMP) will be measured using both TTE and TEE.
Tricuspid annular plane systolic excursion (TAPSE) | Immediately following the induction of anesthesia and TEE probe placement
  Tricuspid annular plane systolic excursion (TAPSE) will be measured using both TTE and TEE.
Right ventricular fractional area change (FAC) | Immediately following the induction of anesthesia and TEE probe placement
  Right ventricular fractional area change (FAC) will be measured using both TTE and TEE.
RV annular systolic velocity (S') | Immediately following the induction of anesthesia and TEE probe placement
  RV annular systolic velocity (S') will be measured using both TTE and TEE.
RV free wall longitudinal strain | Immediately following the induction of anesthesia and TEE probe placement
  RV free wall longitudinal strain will be measured using both TTE and TEE.

SECONDARY OUTCOMES:
Ease of obtaining appropriate TEE measures of right ventricular function | Within 15 minutes following anesthesia induction
  Ease of acquisition will be assessed by the echocardiographers
Define values for normal right ventricular free wall strain | Through study completion, an estimate of 1 year
  The data collected will be used to define normal values for right ventricular free wall strain

CONTACTS AND LOCATIONS:
Overall Officials: Shayne M Roberts, DO, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barakat AF, Sperry BW, Starling RC, Mentias A, Popovic ZB, Griffin BP, Desai MY. Prognostic Utility of Right Ventricular Free Wall Strain in Low Risk Patients After Orthotopic Heart Transplantation. Am J Cardiol. 2017 Jun 1;119(11):1890-1896. doi: 10.1016/j.amjcard.2017.03.003. Epub 2017 Mar 15. PMID 28390683
- [Background] Bellavia D, Iacovoni A, Scardulla C, Moja L, Pilato M, Kushwaha SS, Senni M, Clemenza F, Agnese V, Falletta C, Romano G, Maalouf J, Dandel M. Prediction of right ventricular failure after ventricular assist device implant: systematic review and meta-analysis of observational studies. Eur J Heart Fail. 2017 Jul;19(7):926-946. doi: 10.1002/ejhf.733. Epub 2017 Mar 31. PMID 28371221
- [Background] Howard-Quijano K, Salem A, Barkulis C, Mazor E, Scovotti JC, Ho JK, Shemin RJ, Grogan T, Elashoff D, Mahajan A. Preoperative Three-Dimensional Strain Imaging Identifies Reduction in Left Ventricular Function and Predicts Outcomes After Cardiac Surgery. Anesth Analg. 2017 Feb;124(2):419-428. doi: 10.1213/ANE.0000000000001440. PMID 27782943
- [Background] Kemal HS, Kayikcioglu M, Kultursay H, Vuran O, Nalbantgil S, Mogulkoc N, Can L. Right ventricular free-wall longitudinal speckle tracking strain in patients with pulmonary arterial hypertension under specific treatment. Echocardiography. 2017 Apr;34(4):530-536. doi: 10.1111/echo.13472. Epub 2017 Mar 23. PMID 28332221
- [Background] Peyrou J, Chauvel C, Pathak A, Simon M, Dehant P, Abergel E. Preoperative right ventricular dysfunction is a strong predictor of 3 years survival after cardiac surgery. Clin Res Cardiol. 2017 Sep;106(9):734-742. doi: 10.1007/s00392-017-1117-y. Epub 2017 Apr 13. PMID 28409231
- [Background] Sokalskis V, Peluso D, Jagodzinski A, Sinning C. Added clinical value of applying myocardial deformation imaging to assess right ventricular function. Echocardiography. 2017 Jun;34(6):919-927. doi: 10.1111/echo.13521. Epub 2017 Mar 19. PMID 28317170
- [Background] Tousignant C, Desmet M, Bowry R, Harrington AM, Cruz JD, Mazer CD. Speckle tracking for the intraoperative assessment of right ventricular function: a feasibility study. J Cardiothorac Vasc Anesth. 2010 Apr;24(2):275-9. doi: 10.1053/j.jvca.2009.10.022. Epub 2010 Jan 6. PMID 20056440
- [Background] Agac MT, Akyuz AR, Acar Z, Akdemir R, Korkmaz L, Kiris A, Erkus E, Erkan H, Celik S. Evaluation of right ventricular function in early period following transcatheter closure of atrial septal defect. Echocardiography. 2012 Mar;29(3):358-62. doi: 10.1111/j.1540-8175.2011.01558.x. Epub 2011 Nov 8. PMID 22066780
- [Background] Akiyama K, Arisawa S, Ide M, Iwaya M, Naito Y. Intraoperative cardiac assessment with transesophageal echocardiography for decision-making in cardiac anesthesia. Gen Thorac Cardiovasc Surg. 2013 Jun;61(6):320-9. doi: 10.1007/s11748-013-0208-6. Epub 2013 Feb 13. PMID 23404310
- [Background] Carerj S, Micari A, Trono A, Giordano G, Cerrito M, Zito C, Luzza F, Coglitore S, Arrigo F, Oreto G. Anatomical M-mode: an old-new technique. Echocardiography. 2003 May;20(4):357-61. doi: 10.1046/j.1540-8175.2003.03041.x. PMID 12848879
- [Background] Chan J, Wahi S, Cain P, Marwick TH. Anatomical M-mode: A novel technique for the quantitative evaluation of regional wall motion analysis during dobutamine echocardiography. Int J Card Imaging. 2000 Aug;16(4):247-55. doi: 10.1023/a:1026539708034. PMID 11219596
- [Background] David JS, Tousignant CP, Bowry R. Tricuspid annular velocity in patients undergoing cardiac operation using transesophageal echocardiography. J Am Soc Echocardiogr. 2006 Mar;19(3):329-34. doi: 10.1016/j.echo.2005.09.013. PMID 16500497
- [Background] Hahn RT, Abraham T, Adams MS, Bruce CJ, Glas KE, Lang RM, Reeves ST, Shanewise JS, Siu SC, Stewart W, Picard MH. Guidelines for performing a comprehensive transesophageal echocardiographic examination: recommendations from the American Society of Echocardiography and the Society of Cardiovascular Anesthesiologists. J Am Soc Echocardiogr. 2013 Sep;26(9):921-64. doi: 10.1016/j.echo.2013.07.009. No abstract available. PMID 23998692
- [Background] Ito S, Pislaru SV, Soo WM, Huang R, Greason KL, Mathew V, Sandhu GS, Eleid MF, Suri RM, Oh JK, Nkomo VT. Impact of right ventricular size and function on survival following transcatheter aortic valve replacement. Int J Cardiol. 2016 Oct 15;221:269-74. doi: 10.1016/j.ijcard.2016.07.085. Epub 2016 Jul 6. PMID 27404688
- [Background] Magunia H, Schmid E, Hilberath JN, Haberle L, Grasshoff C, Schlensak C, Rosenberger P, Nowak-Machen M. 2D Echocardiographic Evaluation of Right Ventricular Function Correlates With 3D Volumetric Models in Cardiac Surgery Patients. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):595-601. doi: 10.1053/j.jvca.2016.11.020. Epub 2016 Nov 14. PMID 28129939
- [Background] Markin NW, Chamsi-Pasha M, Luo J, Thomas WR, Brakke TR, Porter TR, Shillcutt SK. Transesophageal Speckle-Tracking Echocardiography Improves Right Ventricular Systolic Function Assessment in the Perioperative Setting. J Am Soc Echocardiogr. 2017 Feb;30(2):180-188. doi: 10.1016/j.echo.2016.10.002. Epub 2016 Dec 1. PMID 27916237
- [Background] Mishra M, Swaminathan M, Malhotra R, Mishra A, Trehan N. Evaluation of Right Ventricular Function During CABG: Transesophageal Echocardiographic Assessment of Hepatic Venous Flow Versus Conventional Right Ventricular Performance Indices. Echocardiography. 1998 Jan;15(1):51-58. doi: 10.1111/j.1540-8175.1998.tb00577.x. PMID 11175010
- [Background] Morita Y, Nomoto K, Fischer GW. Modified Tricuspid Annular Plane Systolic Excursion Using Transesophageal Echocardiography for Assessment of Right Ventricular Function. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):122-6. doi: 10.1053/j.jvca.2015.07.024. Epub 2015 Jul 28. PMID 26520027
- [Background] Niimi Y, Hiki M, Ishiguro Y, Goto T, Morita S. Determination of right ventricular function by transesophageal echocardiography: impact of proximal right coronary artery stenosis. J Clin Anesth. 2004 Mar;16(2):104-10. doi: 10.1016/j.jclinane.2003.05.009. PMID 15110371
- [Background] Portnoy SG, Rudski LG. Echocardiographic evaluation of the right ventricle: a 2014 perspective. Curr Cardiol Rep. 2015;17(4):21. doi: 10.1007/s11886-015-0578-8. PMID 25725606
- [Background] Rafferty T, Durkin M, Harris S, Elefteriades J, Hines R, Prokop E, O'Connor T. Transesophageal two-dimensional echocardiographic analysis of right ventricular systolic performance indices during coronary artery bypass grafting. J Cardiothorac Vasc Anesth. 1993 Apr;7(2):160-6. doi: 10.1016/1053-0770(93)90210-c. PMID 8477020
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Shillcutt SK, Brakke TR, Thomas WR, Porter TR, Lisco SJ. The development of a perioperative echocardiography consult service: the Nebraska experience. J Cardiothorac Vasc Anesth. 2015;29(3):777-84. doi: 10.1053/j.jvca.2014.09.010. Epub 2015 Jan 6. No abstract available. PMID 25575406
- [Background] Shillcutt SK, Markin NW, Montzingo CR, Brakke TR. Use of rapid "rescue" perioperative echocardiography to improve outcomes after hemodynamic instability in noncardiac surgical patients. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):362-70. doi: 10.1053/j.jvca.2011.09.029. Epub 2012 Jan 4. PMID 22226417
- [Background] Strotmann JM, Kvitting JP, Wilkenshoff UM, Wranne B, Hatle L, Sutherland GR. Anatomic M-mode echocardiography: A new approach to assess regional myocardial function--A comparative in vivo and in vitro study of both fundamental and second harmonic imaging modes. J Am Soc Echocardiogr. 1999 May;12(5):300-7. doi: 10.1016/s0894-7317(99)70050-7. PMID 10231615
- [Background] Tousignant C, Bowry R, Cruz JD, Mazer CD. Induction of anesthesia does not alter tricuspid annular velocities: a tissue Doppler assessment. Can J Anaesth. 2009 Oct;56(10):757-62. doi: 10.1007/s12630-009-9157-z. Epub 2009 Jul 29. PMID 19639373
- [Background] Tousignant C, Kim H, Papa F, Mazer CD. Evaluation of TAPSE as a measure of right ventricular output. Can J Anaesth. 2012 Apr;59(4):376-83. doi: 10.1007/s12630-011-9659-3. PMID 22302303
- [Background] Williams B, Sikorski R, Anders M, Galvagno S, Rock P, Mazzeffi M. Should We Use Perioperative Transesophageal Echocardiography More in Non-Cardiac Surgery? J Cardiothorac Vasc Anesth. 2018 Jun;32(3):e71-e73. doi: 10.1053/j.jvca.2016.03.153. Epub 2016 Mar 31. No abstract available. PMID 27474334